CLINICAL TRIAL: NCT02866565
Title: Assessment of the Efficacy and Tolerance of Sub-cutaneous Re-injection of Autologous
Brief Title: Assessment of the Efficacy and Tolerance of Sub-cutaneous Re-injection of Autologous Adipose-derived REGEnerative Cells in the Local Treatment of Neuropathic Diabetic Foot ulcERs
Acronym: REGENDER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-41
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetic foot ulcer (Experimental)
  Interventions: Drug: adipose-derived regenerative cells (ADRCs)

INTERVENTIONS:
Drug: adipose-derived regenerative cells (ADRCs) — injection of the experimental treatment

SUMMARY:
Diabetic foot ulcer (DFU) is a major complication and the leading cause of hospitalization among people with diabetes mellitus. It occurs in 15% of all patients with diabetes and precedes 84% of all lower leg amputations. Despite many therapeutic advances over the past decades, including dressings (hydrocolloids, alginate, skin substitutes) and growth factors, healing rates of DFU remain low.

Mechanisms of faulty wound healing in diabetic patients are complex, related to both intrinsic and extrinsic factors. The main reasons for impaired healing appears to be: 1/exhaustion of local cell populations that promote wound healing; 2/excessive production of matrix metalloproteases (MMPs) coupled with reduced expression of the tissue inhibitors of MMPs; 3/impaired neovascularisation coupled with reduced numbers of endothelial progenitor cells and impairment of their functioning. These imbalances may result in excessive degradation of extracellular matrix components, as well as an inappropriate local inflammatory response .

Adipose-derived stroma vascular fraction provides a rich and easily accessible source of autologous cells for regenerative medicine applications. Il contains multipotent stem cells and progenitors called adipose-derived regenerative cells (ADRCs) able to stimulate wound healing. There are attracted to the wound site where they supplement the wound bed with similar cell types, secrete numerous growth factors and cytokines, increase macrophage recruitment, enhance granulation tissue, and improve vascularisation . The reparative capabilities coupled with good safety of ADRCs have been illustrated in a study for treating severe and irreversible radiation-induced lesions, and in a study for treating sclerodactyly in patients with diffuse scleroderma. Numerous case reports showing healing of refractory wounds following treatment with autologous ADRCs have also been reported.

Based on these previous reports, the present study aims to assess the efficacy and tolerance of injection of ADRCs for the local treatment of neuropathic or neuro-ischemic DFU.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18
* Patient with type 1 or 2 diabetes mellitus with HbA1C level < 10%
* Patient with diagnosis of neuropathic or neuro-ischemic DFU
* Grade 1 or 2 ulcer on the Wagner scale
* Ulcer with a surface area comprised between 1 cm2 and 15 cm2 at day 0 Patient present for a minimum of 4 weeks under the current investigator's care including adequate wound debridement and offloading
* Semmes-Weinstein monofilament test indicating neuropathy
* DFU located on the toe or on the lateral, dorsal surface of the forefoot or heel

Exclusion Criteria:

* Pregnant or likely to become pregnant or breast feeding woman
* Critical ischemia of the target limb, defined by pain at rest and an ankle systolic pressure < 50 mm Hg, or a toe systolic pressure < 30 mm Hg
* Surgery or surgical revascularisation < 2months
* Decrease or increase in the ulcer size by 30% or more within a 2-wk run-in period
* DFU clinically infected as defined by the IDSA/IWGDF criteria, osteomyelitis confirmed by MRI, or other evidence of infection is present Dossier LIC-15-15-0005 REGENDER Déposé le 09/03/2015 15:22:11 par M. Patrice DARMON Appel LIC-15-2015 Page 3 sur 6
* Patient who cannot bear an off-loading method
* Patient with an active neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving 100% wound closure | 20 WEEKS

SECONDARY OUTCOMES:
time to reach complete wound closure | 20 WEEKS
wound surface regression in relative value | 20 weeks
wound surface regression in absolute value | 20 weeks
percentage of patients achieving 50 % wound closure | 20 weeks
ulcer recurrence rate | 20 weeks
change in quality of life assessed by the SF-36 QoL survey from baseline | 20weeks

CONTACTS AND LOCATIONS:
Overall Officials: catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille; PATRICE DARMON, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France